CLINICAL TRIAL: NCT04686305
Title: A Phase Ib Multicenter, Open-label Study to Evaluate the Safety and Tolerability of Trastuzumab Deruxtecan (T-DXd) and Immunotherapy Agents With and Without Chemotherapy Agents in First-line Treatment of Patients With Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer (NSCLC) and Human Epidermal Growth Factor Receptor 2 (HER2) Overexpression (OE) (DESTINY-Lung03)
Brief Title: Phase Ib Study of the Safety of T-DXd and Immunotherapy Agents With and Without Chemotherapy in Advanced or Metastatic HER2+, Non-squamous NSCLC
Acronym: DL03
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D967YC00001; 2023-504949-31-00 (Registry Identifier: CTIS); 2020-003260-31 (EudraCT Number)
Record Dates: First submitted 2020-12-08; First posted 2020-12-28 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Keywords: HER2+; HER2 expression; DS-8201a; T-DXd; Trastuzumab Deruxtecan; Volrustomig (MEDI5752); Antibody - drug conjugate; bispecific antibody; Volrustomig; Rilvegostomig; Carboplatin; First line; Locally advanced and unresectable non-squamous NSCLC; Metastatic non-squamous NSCLC; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — trastuzumab deruxtecan; durvalumab; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: DL-03 aims to identify T-DXd-based combination therapies for patients with previously untreated, advanced, HER2-overexpressing NSCLC. Across all study parts, the primary objectives are to assess safety and tolerability. Secondary objectives include assessing preliminary efficacy based on ORR, DoR, DCR, PFS, and OS. Part 5 will consist of two arms evaluating T-DXd plus volrustomig, without chemotherapy. Arm 5A will assess T-DXd plus volrustomig as a single priming dose, followed by a lower, fixed maintenance dose. Arm 5B will evaluate T-DXd plus volrustomig as fixed doses. Part 4 consists of two arms utilizing T-DXd plus rilvegostomig, without or with carboplatin (first 4 cycles in Arm 4B only). Part 3 consists of two arms utilizing T-DXd plus volrustomig, without or with carboplatin (first 4 cycles in Arm 3B only), and assesses two different volrustomig doses. Part 3 is closed to recruitment and enrolment. Part 2 was not initiated. Part 1 is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Arm 1A: T-DXd, Durvalumab and Cisplatin (Experimental): T-DXd, Durvalumab and Cisplatin
  Interventions: Drug: T-DXd; Biological: Durvalumab; Drug: Cisplatin
- Arm 1B: T-DXd, Durvalumab and Carboplatin (Experimental): T-DXd, Durvalumab and Carboplatin
  Interventions: Drug: T-DXd; Biological: Durvalumab; Drug: Carboplatin
- Arm 1C: T-DXd, Durvalumab and Pemetrexed (Experimental): T-DXd, Durvalumab and Pemetrexed (Arm not initiated)
  Interventions: Drug: T-DXd; Biological: Durvalumab; Drug: Pemetrexed
- Arm 1D: T-DXd (Experimental): T-DXd
  Interventions: Drug: T-DXd
- Arm 3A: T-DXd and Volrustomig (Experimental): Drug: T-DXd and Volrustomig T-DXd: administered as an IV infusion Other Name: DS-8201a, Trastuzumab deruxtecan Biological/Vaccine: Volrustomig Volrustomig: administered as an IV infusion Other Name: Volrustomig
  Interventions: Drug: T-DXd; Drug: Volrustomig
- Arm 3B: T-DXd, Volrustomig and Carboplatin (Experimental): Drug: T-DXd, Volrustomig and Carboplatin T-DXd: administered as an IV infusion Other Name: DS-8201a, Trastuzumab deruxtecan Biological/Vaccine: Volrustomig Volrustomig: administered as an IV infusion Other Name: Volrustomig Drug: Carboplatin Carboplatin: administered as an IV infusion
  Interventions: Drug: T-DXd; Drug: Carboplatin; Drug: Volrustomig
- Arm 4A: T-DXd and Rilvegostomig (Experimental): T-DXd and Rilvegostomig Drug: T-DXd, Rilvegostomig T-DXd: administered as an IV infusion Other Name: DS-8201a, Trastuzumab deruxtecan Biological/Vaccine: Rilvegostomig Rilvegostomig: administered as an IV infusion Other Name: Rilvegostomig, AZD2936
  Interventions: Drug: T-DXd; Drug: Rilvegostomig
- Arm 4B T-DXd and Rilvegostomig with Carboplatin (Experimental): Drug: T-DXd, Rilvegostomig and Carboplatin T-DXd: administered as an IV infusion Other Name: DS-8201a, Trastuzumab deruxtecan Biological/Vaccine: Rilvegostomig Rilvegostomig: administered as an IV infusion Other Name: Rilvegostomig, AZD2936 Drug: Carboplatin Carboplatin: administered as an IV infusion
  Interventions: Drug: T-DXd; Drug: Carboplatin; Drug: Rilvegostomig
- Arm 5A: T-DXd and Volrustomig (Experimental): Drug: T-DXd and volrustomig T-DXd: administered as an IV infusion Other Name: DS-8201a, trastuzumab deruxtecan Biological/Vaccine: Volrustomig Volrustomig: administered as an IV infusion (priming dose in first cycle, fixed dose in subsequent cycles) Other Name: volrustomig
  Interventions: Drug: T-DXd; Drug: Volrustomig
- Arm 5B: T-DXd and Volrustomig (Experimental): Drug: T-DXd and volrustomig T-DXd: administered as an IV infusion Other Name: DS-8201a, trastuzumab deruxtecan Biological/Vaccine: Volrustomig Volrustomig: administered as an IV infusion (fixed dose from first cycle onward) Other Name: volrustomig
  Interventions: Drug: T-DXd; Drug: Volrustomig

INTERVENTIONS:
Drug: T-DXd — T-DXd: administered as an IV infusion
  Other Names: DS-8201a, Trastuzumab deruxtecan
Biological: Durvalumab — Durvalumab: administered as an IV infusion
  Other Names: MEDI4736
  Arms: Arm 1A: T-DXd, Durvalumab and Cisplatin; Arm 1B: T-DXd, Durvalumab and Carboplatin; Arm 1C: T-DXd, Durvalumab and Pemetrexed
Drug: Cisplatin — Cisplatin: administered as an IV infusion
  Arms: Arm 1A: T-DXd, Durvalumab and Cisplatin
Drug: Carboplatin — Carboplatin: administered as an IV infusion
  Arms: Arm 1B: T-DXd, Durvalumab and Carboplatin; Arm 3B: T-DXd, Volrustomig and Carboplatin; Arm 4B T-DXd and Rilvegostomig with Carboplatin
Drug: Pemetrexed — Pemetrexed: administered as an IV infusion (drug not used)
  Arms: Arm 1C: T-DXd, Durvalumab and Pemetrexed
Drug: Volrustomig — Volrustomig: administered as an IV infusion
  Other Names: Other Name: MEDI5752
  Arms: Arm 3A: T-DXd and Volrustomig; Arm 3B: T-DXd, Volrustomig and Carboplatin; Arm 5A: T-DXd and Volrustomig; Arm 5B: T-DXd and Volrustomig
Drug: Rilvegostomig — Rilvegostomig: administered as an IV infusion
  Other Names: Other Name: AZD2936
  Arms: Arm 4A: T-DXd and Rilvegostomig; Arm 4B T-DXd and Rilvegostomig with Carboplatin

SUMMARY:
DESTINY-Lung03 will investigate the safety and tolerability of trastuzumab deruxtecan in combination with Immunotherapy Agents with and without chemotherapy in patients with HER2 over-expressing non-small cell lung cancer. The efficacy will be also analyzed as a secondary endpoint.

DETAILED DESCRIPTION:
Part 1 is a dose escalation study by design, allowing the assessment of safety, tolerability, and recommended dose levels of the combination of T-DXd and durvalumab plus cisplatin, carboplatin, or pemetrexed. No more patients will be enrolled in this part of the study. Part 2, expansions in the treatment-naïve setting on any recommended dose level, will not be initiated.

The evaluation of T-DXd combination treatment with immunotherapy continues in Part 3, Part 4, and Part 5. In Part 3, T-DXd is assessed in combination with volrustomig, with carboplatin (Arm 3B) or without carboplatin (Arm 3A). Part 4 examines T-DXd with rilvegostomig, either with carboplatin (Arm 4B) or without carboplatin (Arm 4A). In Part 5, T-DXd is evaluated with volrustomig, given with or without a priming dose followed by a fixed dose in Arm 5A. There is also an optional Arm 5B at the Sponsor's discretion. These parts focus on further dose optimization for first-line HER2-overexpressing NSCLC.

For Part 3, patients will be randomized to Arms 3A and 3B, beginning with the cohorts receiving the volrustomig starting dose (SD). A total of 6 DLT-evaluable patients will be enrolled to the SD cohorts in each arm. If the combination of T-DXd with volrustomig at the starting dose is deemed safe, a dose escalation (E1) cohort will be opened for 6 DLT-evaluable patients. Once all open dose confirmation cohorts have 6 DLT-evaluable patients, the SRC will convene to select the volrustomig RP2D to be used in the dose-expansion (DE) cohorts of each arm (n=34). Part 3 is now permanently closed to recruitment; no further patients will be enrolled.

In Part 4, once a total of 6 DLT-evaluable patients/arm have been enrolled into Arm 4A and Arm 4B safety-run in (SR) cohorts and deemed safe, an additional 34 patients per arm will be enrolled in Arms 4A and 4B in dose expansion cohorts.

Part 5 involves additional dosing regimens of T-DXd in combination with volrustomig. The objective of Part 5 is to evaluate the safety and efficacy of priming and flat dosing regimens in 2 different cohorts of up to 30 patients per arm.

The target population of interest (for Part 3, 4 and 5) are patients with advanced or metastatic non-small cell lung cancer measurable disease by RECIST 1.1 criteria, HER2 overexpression, ECOG PS of 0 to 1, patients who are treatment naïve for recurrent, unresectable or metastatic disease. Patients with tumors that harbor a known genomic alteration or driver for which approved therapies are available are excluded.

ELIGIBILITY:
Inclusion criteria:

* Histologically documented unresectable locally advanced/metastatic non-squamous NSCLC
* Part 1: Progression after 1 or 2 lines of systemic therapy for recurrent or metastatic setting.
* Part 3, Part 4 and Part 5: Patients must have tumors that do not harbor known genomic alterations or actionable driver kinases, for which approved therapies are available are allowed.
* Part 3, Part 4 and Part 5: Patient must be treatment-naïve for advanced or metastatic NSCLC. Patients who have received prior adjuvant, or neoadjuvant chemotherapy, or definitive chemoradiation for advanced disease are eligible, provided that progression has occurred > 6 months from end of last therapy
* HER2overexpression status as determined by central review of tumor tissue
* WHO / ECOG performance status of 0 or 1
* Measurable target disease assessed by the investigator using RECIST 1.1
* Has protocol defined adequate organ and bone marrow function
* Part 3, Part 4 and Part 5: Minimum body weight of 35 kg.

Exclusion criteria:

* HER2 mutation if previously known
* Has a history of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder and prior pneumonectomy
* Active primary immunodeficiency known HIV infection, or active chronic and resolved hepatitis B (positive hepatitis B virus surface antigen [HBsAg+ve] or hepatitis B virus core antibody (anti-HBc +ve) regardless of HBV DNA level)) or hepatitis C infection. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Patients should be tested for HIV prior to treatment assignment if required by local regulations or IRB/EC
* Active infection including tuberculosis and uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
* Spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms
* Medical history of myocardial infarction within 6 months before treatment assignment, symptomatic CHF (New York Heart Association Class II to IV), clinically important cardiac arrhythmias, or a recent (< 6 months) cardiovascular event including stroke
* For Part 3, Part 4 and Part 5: Cardiomyopathy of any etiology, symptomatic CHF (as defined by New York Heart Association Class > II), unstable angina pectoris, history of MI within the past 12 months, or cardiac arrhythmia are to be excluded. Patients with troponin levels above ULN at screening (as defined by the manufacturer), and without any myocardial related symptoms, should have a cardiologic consultation before treatment assignment to rule out acute cardiopulmonary events.
* Ascites or pericardial effusion that requires drainage, peritoneal shunt, Pleuroperitoneal shunt or CART (Concentrated Ascites Reinfusion Therapy)
* For Part 3, Part 4 and Part 5: Active non-infectious skin disease (including any grade rash, urticarial, dermatitis, ulceration, or psoriasis) requiring systemic treatment, active or prior documented autoimmune or inflammatory disorders requiring chronic treatment with steroids or other immunosuppressive treatment.
* Unresolved toxicities not yet resolved to Grade ≤ 1 or baseline from previous anticancer therapy OR prior discontinuation of any planned study therapy due to toxicity.
* must not have any medical contraindication to platinum-based chemotherapy.
* Part 3, Part 4 and Part 5 patients must not have had prior exposure to anti-PD-1, anti-PD-L1, anti-CTLA-4, anti-TIGIT or any other experimental immunotherapy in any setting.
* For Part 3, Part 4 and Part 5: History of substance abuse or any other medical or psychological conditions that may, in the opinion of the Investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results
* For Part 3, Part 4 and Part 5: History of thromboembolic events within 3 months before the first dose of IP (limited to pulmonary embolism, deep vein thrombosis, or cerebral venous sinus thrombosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of AEs and SAEs | Safety and tolerability (and to determine RP2D) will be assessed for approximately 20 months from informed consent
  Occurrence of AEs and SAEs graded according to NCI CTCAE v5.0

SECONDARY OUTCOMES:
Confirmed Objective Response Rate (ORR) | An average of approximately 12 months
  Confirmed ORR per RECIST 1.1 is the percentage of patients with Complete Response or Partial Response that is subsequently confirmed, based on investigator assessment
Duration of Response (DoR) | An average of approximately 20 months
  DOR is defined as the time from the date of first documented response until the date of documented progression or death, based on RECIST 1.1 assessment
Disease Control Rate (DCR) | An average of approximately 12 months
  DCR is the percentage of patients who have a best overall response of complete response (CR) or partial response (PR) or stable disease (SD), based on RECIST 1.1 assessment. DCR is assessed at 6 and 12 weeks
Progression-free survival (PFS) | An average of approximately 20 months
  PFS is the time from first dose of study treatment until the date of objective disease progression or death, based on RECIST 1.1 assessment
Overall survival (OS) | An average of approximately 20 months
  OS is the time form the date of first dose of study treatment until death due to any cause
Pharmacokinetics (PK) assessed by the serum concentration of T-DXd, total anti-HER2 antibody, and MAAA-1181 in all arms | An average of approximately 20 months
  Individual patient data and descriptive statistics will be provided for serum concentration data at each time point for T-DXd, total anti-HER2 antibody and MAAA-1181a
Pharmacokinetics (PK) assessed by the serum concentration of durvalumab in study arms including T-DXd in combination with durvalumab | An average of approximately 20 months
  Individual patient data and descriptive statistics will be provided for serum concentration data at each time point for durvalumab, including T-DXd in combination with durvalumab
Pharmacokinetics (PK) assessed by the serum concentration of volrustomig in study arms including T-DXd in combination with volrustomig | An average of approximately 20 months
  Individual patient data and descriptive statistics will be provided for serum concentration data at each time point for volrustomig, including T-DXd in combination with volrustomig
Pharmacokinetics (PK) assessed by the serum concentration of rilvegostomig in study arms including T-DXd in combination with rilvegostomig | An average of approximately 20 months
  Individual patient data and descriptive statistics will be provided for serum concentration data at each time point for rilvegostomig, including T- DXd in combination with rilvegostomig
The immunogenicity of T-DXd, durvalumab, volrustomig and rilvegostomig assessed by the presence of ADAs for T-DXd, durvalumab, volrustomig, or rilvegostomig | An average of approximately 20 months
  Individual participant data and descriptive statistics will be provided for data at each time point for each dose level for T-DXd, durvalumab or volrustomig, or rilvegostomig

CONTACTS AND LOCATIONS:
Locations (73):
- United States (13):
  - Research Site, Duarte, California
  - Research Site, Newport Beach, California
  - Research Site, Orange, California
  - Research Site, Santa Rosa, California
  - Research Site, Westwood, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Tacoma, Washington
- Australia (3):
  - Research Site, Adelaide
  - Research Site, Heidelberg
  - Research Site, Nedlands
- Research Site, Edegem, Belgium
- Brazil (3):
  - Research Site, Barretos
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Canada (3):
  - Research Site, Winnipeg, Manitoba
  - Research Site, London, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Fuzhou, China
- France (5):
  - Research Site, Bordeaux
  - Research Site, Dijon
  - Research Site, Pierre-Bénite
  - Research Site, Saint-Herblain
  - Research Site, Villejuif
- Israel (2):
  - Research Site, Kfar Saba
  - Research Site, Tel Litwinsky
- Italy (4):
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Padua
- Malaysia (4):
  - Research Site, George Town
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Kuching
- Research Site, Amsterdam, Netherlands
- Philippines (7):
  - Research Site, Bacolod
  - Research Site, Cebu City
  - Research Site, City of Taguig
  - Research Site, Davao City
  - Research Site, Manila
  - Research Site, Quezon City
  - Research Site, San Juan City
- Poland (5):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Olsztyn
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
- Research Site, Singapore, Singapore
- South Korea (4):
  - Research Site, Cheongju-si
  - Research Site, Goyang-si
  - Research Site, Jinju
  - Research Site, Seoul
- Spain (4):
  - Research Site, Badalona
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Bornova-Izmir
  - Research Site, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Planchard D, Kim HR, Suksombooncharoen T, Li R, Cortinovis D, Han JY, Samol J, Runglodvatana Y, Lee KY, Chang GC, Lee CH, Kowalski D, Saw SPL, Huang Y, Ruiter G, Ahn MJ, Yang TY, Yang CT, Sookprasert A, Nakajima EC, Alfon J, McEwen R, Chang YT, Yang JC. Trastuzumab Deruxtecan in Patients With HER2-Overexpressing NSCLC: Results From Part 1 of the Open-Label, Multicenter, Phase 1b DESTINY-Lung03 Trial. J Thorac Oncol. 2025 Dec 23:103541. doi: 10.1016/j.jtho.2025.12.080. Online ahead of print. PMID 41448488
- See also: Lung Cancer Study Locator details (for US) — https://www.lungcancerstudylocator.com/trial/listing/264517